CLINICAL TRIAL: NCT00415116
Title: Phase I Trial of Three-Weekly Docetaxel, Carboplatin and Oral CC-5013 in Patients With Advanced Solid Tumors
Brief Title: Lenalidomide, Docetaxel, and Carboplatin in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Tarek Mekhail, Cleveland Clinic Taussing Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE-CCF-7216; P30CA043703 (NIH); CASE-CCF-7216
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2006-11

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Carboplatin; Docetaxel; Lenalidomide

INTERVENTIONS:
Drug: carboplatin
Drug: docetaxel
Drug: lenalidomide

SUMMARY:
RATIONALE: Lenalidomide may stop the growth of solid tumors by blocking blood flow to the tumor. Drugs used in chemotherapy, such as docetaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving lenalidomide together with docetaxel and carboplatin may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of lenalidomide when given together with docetaxel and carboplatin in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of lenalidomide when administered with docetaxel and carboplatin in patients with advanced solid tumors.

Secondary

* Determine the safety and toxic effects of this regimen in these patients.
* Determine, preliminarily, the clinical activity of this regimen in these patients.

OUTLINE: This is an open-label, dose-escalation study of lenalidomide.

Patients receive docetaxel IV over 1 hour followed by carboplatin IV on day 1. Patients also receive oral lenalidomide once daily on days 1-14. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease after completion of 6 courses of treatment may continue lenalidomide alone once daily on days 1-14. Patients whose disease is stable or responding after completing 2 or 4 courses and who are unable to tolerate further chemotherapy may continue lenalidomide alone once daily on days 1-14, at the investigator's discretion. Treatment with lenalidomide repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of lenalidomide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. An additional 6-8 patients are treated at the MTD.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven solid tumor
* Measurable or evaluable disease
* Refractory to standard treatment
* No prior failure of a docetaxel and carboplatin regimen except in the adjuvant setting
* History of brain disease allowed, provided the following criteria are met:

  * Brain disease previously treated with radiotherapy or surgery
  * Asymptomatic with no active brain disease, as documented by CT scan or MRI, for at least 3 months

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 1.5 mg/dL
* Bilirubin normal
* AST and ALT ≤ 2 times upper limit of normal (ULN) (5 times ULN if hepatic metastases are present)
* Alkaline phosphatase ≤ 3 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 weeks after completion of study treatment
* No serious medical condition, laboratory abnormality, or psychiatric illness that would preclude giving informed consent, expose the patient to unacceptable risk, or affect the interpretation of study data
* No known hypersensitivity to thalidomide
* No history of erythema nodosum, characterized by a desquamating rash, while taking thalidomide or similar drugs
* No pre-existing peripheral neuropathy ≥ grade 2
* No known hypersensitivity or intolerance to taxanes
* No known HIV positivity
* No known infectious hepatitis, types A, B, or C

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than 2 prior chemotherapy regimens
* At least 28 days since prior cancer therapy, including radiotherapy, biologic therapy, hormonal therapy, chemotherapy, or surgery
* At least 28 days since any other prior investigational drug or therapy
* No prior lenalidomide
* No other concurrent chemotherapy or biologic therapy
* No concurrent radiotherapy
* No concurrent use of any other anticancer agents or treatments
* No prophylactic granulocyte colony-stimulating factors (G-CSF) during the first course of study treatment
* No concurrent prophylactic antibiotics
* No concurrent treatment with the following medications:

  * Systemic corticosteroids (except as prophylaxis for docetaxel administration)
  * Estrogens
  * Azoles
  * Macrolides
  * Cyclosporine
  * Rifampin
  * Phenytoin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2004-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of lenalidomide
Dose-limiting toxicity of lenalidomide

SECONDARY OUTCOMES:
Safety and toxicity
Clinical activity

CONTACTS AND LOCATIONS:
Overall Officials: Tarek M. Mekhail, MD, Study Chair — Case Comprehensive Cancer Center